CLINICAL TRIAL: NCT01364233
Title: A Prospective Outcome Study of Condensed Fenestrated PTFE Mesh (MotifMESH) in Non-sterile Abdominal Wall Defects
Brief Title: Safety Study of MotifMESH (cPTFE) in Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-NU-2011-01
Record Dates: First submitted 2011-05-27; First posted 2011-06-02 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MotifMesh (Other): Condensed polytetrafluoroethylene (cPTFE, MotifMESH) mesh
  Interventions: Device: MotifMESH

INTERVENTIONS:
Device: MotifMESH — Polytetrafluoroethylene (cPTFE) macroporous mesh

SUMMARY:
This study will monitor surgically repaired large abdominal hernias requiring condensed fenestrated polytetrafluoroethylene mesh (cPTFE).

DETAILED DESCRIPTION:
cPTFEi s a mesh-like product designed to reduce associated post surgical complications.

ELIGIBILITY:
Inclusion Criteria:

Has a non-sterile abdominal wall defect (incisional hernia or fascial defect) and needs to be repaired

Exclusion Criteria:

Non-pregnant, breast feeding or plans to become pregnant during the study; Using adequate birth control methods and agrees to continue using those methods for the duration of the study

Confirmation of incisional hernia or fascial defect by CT scan within 6 months Incisional hernia or facial defect has no necrotic tissue. Such as fascial dehiscence, evisceration, small or large bowel repair, stoma manipulation, small chronic abdominal skin wounds, bowel obstruction

Acceptable state of health and nutrition with pre-albumin levels of ≥ 15 mg/dL (0.15 g/L), serum albumin ≥ 2.0 g/dL (20 g/L). No abnormal pre-surgery laboratory values that, in the opinion of the Principal Investigator, place the subject at risk for the study.

For subjects with Diabetes Mellitus, HbA1C <12%

BMI ≤ 40 kg/m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Dumanian, MD, Principal Investigator — Northwestern University
Locations (1):
- Division of Plastic Surgery, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MotifMesh: Condensed polytetrafluoroethylene (cPTFE, MotifMESH) mesh
  MotifMESH: Polytetrafluoroethylene (cPTFE) macroporous mesh
  MotifMESH: Surgical mesh
Period: Overall Study
Arm/Group | MotifMesh
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- MotifMesh: Participants received Condensed polytetrafluoroethylene (cPTFE, MotifMESH) mesh
Arm/Group | MotifMesh
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Had an Additional Hernia Occur Following Surgery With Condensed Polytetrafluoroethylene (cPTFE, MotifMESH) Mesh
Description: Hernia occurrence at one year after surgery
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Hernia Occurrence at One Year After Surgery: Number of subjects who had an additional hernia occur following surgery with Condensed polytetrafluoroethylene (cPTFE, MotifMESH) mesh post 1 year after initial surgery.
Arm/Group | Hernia Occurrence at One Year After Surgery
Number analyzed (Participants) | 9
participants | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | MotifMesh
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MotifMesh (N=10)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) — Small hematoma located in the lateral incision for performance of a components release, hematoma was drained and resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No